CLINICAL TRIAL: NCT03623243
Title: Exploring the Safety and Tolerability of Conversion From Oral, Injectable, or Infusion Disease Modifying Therapies to Dose-titrated Oral Siponimod (Mayzent) in Patients With Advancing Forms of Relapsing Multiple Sclerosis: A 6-month Open Label, Multi- Center Phase IIIb Study
Brief Title: Safety and Tolerability of Conversion From Oral, Injectable, or Infusion Disease Modifying Therapies to Dose-titrated Oral Siponimod (Mayzent) in Advancing RMS Patients
Acronym: EXCHANGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBAF312AUS02
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis; Relapsing Multiple Sclerosis; Advancing Multiple Sclerosis
Keywords: Multiple sclerosis; Relapsing multiple sclerosis; Advancing multiple sclerosis; conversion; siponimod; adult; BAF312; disease modifying therapies; cognitive assessment; open-label
MeSH Terms: conditions — Multiple Sclerosis | interventions — siponimod

STUDY DESIGN:
Intervention Model Description: Open-label single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Siponimod (Experimental): Participants will receive titrated doses of siponimod tablets, orally, once daily of 0.25 mg on Day 2, 0.5 mg on Day 3, 0.75 mg on Day 4, 1.25 mg on Day 5, and maintenance dose of siponimod 2.0 mg tablets, orally, once daily from Day 6 up to 6 months.
  As of protocol amendment 3, participants entering the trial converting from fingolimod will start directly with 2 mg dose of siponimod.
  Interventions: Drug: Siponimod

INTERVENTIONS:
Drug: Siponimod — Siponimod 2mg tablets taken once daily
  Other Names: BAF312

SUMMARY:
To assess safety and tolerability of patients converting from approved Relapsing Multiple Sclerosis (RMS) Disease Modifying Therapies (DMTs) to siponimod.

DETAILED DESCRIPTION:
This is a 6-month, open-label, multi-center, single arm design, including advancing RMS patients, evaluating the overall safety and tolerability profile of converting from oral, injectable or infusion RMS DMTs to oral siponimod.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed informed consent.
2. Male or female aged 18 to 65 years (inclusive).
3. Patients with advancing RMS as defined by the principal investigator.
4. Prior history of relapsing MS (RMS), with or without progressive features, according to the 2010 Revised McDonald or Lublin criteria (Lublin et al, 2013).
5. EDSS score of >/= 2.0 to 6.5 (inclusive).
6. Having been continuously treated with RMS Disease Modifying Therapies.

Key Exclusion criteria:

1. Pregnant or nursing (lactating) women.
2. Patients with any medically unstable condition as determined by the investigator.
3. Certain cardiac risk factors defined in the protocol
4. History of hypersensitivity to the study drug or to drugs of similar chemical classes.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (53):
- United States (52):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Cullman, Alabama
  - Alabama Neurology Associates, Homewood, Alabama
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Irvine, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Fort Collins, Colorado
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Bradenton, Florida
  - MS & Neuromuscular Center of Excellence, Clearwater, Florida
  - Novartis Investigative Site, Maitland, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Ocala, Florida
  - Novartis Investigative Site, Oldsmar, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Ormond Beach, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Sunrise, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Vero Beach, Florida
  - Novartis Investigative Site, Flossmoor, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, Clinton Township, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Hackensack, New Jersey
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Abington Neurological Associates, Ltd, Abington, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Willow Grove, Pennsylvania
  - Novartis Investigative Site, Greer, South Carolina
  - Novartis Investigative Site, Old Point Station, South Carolina
  - Novartis Investigative Site, Cordova, Tennessee
  - Novartis Investigative Site, Johnson City, Tennessee
  - Novartis Investigative Site, Round Rock, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Falls Church, Virginia
  - Novartis Investigative Site, Kirkland, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Waukesha, Wisconsin
- Novartis Investigative Site, Guaynabo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Fox RJ, Cohan S, Mao-Draayer Y, Weinstock-Guttman B, Cruz LA, Arnould S, Cox GM, Bar-Or A. Safety and tolerability of conversion to siponimod from other disease-modifying therapies in patients with advancing forms of relapsing MS: Results from the EXCHANGE study. Mult Scler. 2025 May;31(6):706-718. doi: 10.1177/13524585251330085. Epub 2025 Apr 18. PMID 40248858
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1555

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States from 14 February 2019 to 06 July 2022.
Pre-assignment Details: A total of 342 participants were screened of which 185 participants were enrolled to receive siponimod.
Groups:
- Siponimod: Participants received titrated doses of siponimod tablets, orally, once daily of 0.25 mg on Day 2, 0.5 mg on Day 3, 0.75 mg on Day 4, 1.25 mg on Day 5, and maintenance dose of siponimod 2.0 mg tablets, orally, once daily from Day 6 up to 6 months.
  As of protocol amendment 3, participants entering the trial converting from fingolimod started directly with 2 mg dose of siponimod.
Period: Overall Study
Arm/Group | Siponimod
Started | 185
Safety Set (Safety set included all participants who received at least one dose of study treatment.) | 185
Completed | 146
Not Completed | 39
Not completed — Adverse Event | 15
Not completed — Guardian Decision | 1
Not completed — New Therapy for Study Indication | 1
Not completed — Protocol Deviation | 3
Not completed — Physician Decision | 4
Not completed — Patient Decision | 15

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received at least one dose of study treatment.
Arm/Group | Siponimod
Number analyzed (Participants) | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39
  Not Hispanic or Latino | 145
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 157
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 185

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE) Related to Study Drug During the Treatment Period
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAEs are defined as the AEs started after the first dose of siponimod to 30 days after the date of the last actual administration, or events present prior to start of treatment but which increased in severity. TEAEs suspected to be related to study drug are reported.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to 7 months)
Population: Safety set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Siponimod
Number analyzed (Participants) | 185
Participants | 59

2. Secondary Outcome: Number of Participants With at Least One Adverse Event (AE)
Description: AE is any untoward sign or symptom that occurs during the study treatment plus 30 days post treatment.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to 7 months)
Population: Safety set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Siponimod
Number analyzed (Participants) | 185
Participants | 138

3. Secondary Outcome: Change From Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM-9)
Description: TSQM-9 measures participant satisfaction with the medication in 3 domains: Effectiveness, convenience, and global satisfaction. The scores were computed by adding items for each domain, i.e., 1 to 3 for effectiveness, 4 to 6 for convenience, and 7 to 9 for global satisfaction. The lowest possible score (1 for each item and 3 for all 3 subscales) was subtracted from the composite score and divided by the greatest possible score range. The greatest range was (7-1) x 3 items = 18 for effectiveness and convenience, and (5-1) x 3 items = 12 for global satisfaction. This provided a transformed score between 0 and 1 that was then multiplied by 100. TSQM-9 domain scores range from 0 to 100, with higher scores indicating greater satisfaction for that domain. A positive change from baseline indicates improvement.
Time Frame: Baseline up to Day 168
Population: Safety set included all participants who received at least one dose of study treatment. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Siponimod
Number analyzed (Participants) | 97
score on a scale
  Change From Baseline in Effectiveness | 13.5 (25.64)
  Change From Baseline in Convenience | 15.6 (25.52)
  Change From Baseline in Global Satisfaction | 15.3 (27.90)

4. Secondary Outcome: Change in Heart Rate From Baseline to 6 Hours After First Treatment
Description: Heart rate was evaluated from the time of initial dose intake until 6 hours post dose intake via heart monitor.
Time Frame: From the first dose up to 6 hours
Population: Safety set included all participants who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Siponimod
Number analyzed (Participants) | 185
beats per minute (bpm) | 2.47 (12.169)

5. Secondary Outcome: Number of Participants With at Least One Hospitalization During the Treatment
Time Frame: From first dose of study drug up to last dose of study drug (up to 6 months)
Population: Safety set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Siponimod
Number analyzed (Participants) | 185
Participants | 9

6. Secondary Outcome: Patient Retention Reported as Number of Participants Who Completed the Study
Description: Patient retention was assessed over the study period.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to 7 months)
Population: Safety set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Siponimod
Number analyzed (Participants) | 185
Participants | 146

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to 7 months)
Description: Safety set included all participants who received at least one dose of study treatment.
Arm/Group | Siponimod
All-Cause Mortality (participants affected / at risk) | 0/185
Serious Adverse Events (participants affected / at risk) | 9/185
Other Adverse Events (participants affected / at risk) | 63/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Siponimod (N=185)
Non-cardiac chest pain (General disorders) | 1
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia aspiration (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Multiple sclerosis (Nervous system disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1
Lymphoedema (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Siponimod (N=185)
Nausea (Gastrointestinal disorders) | 15
Fatigue (General disorders) | 13
Urinary tract infection (Infections and infestations) | 16
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT03623243/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT03623243/SAP_001.pdf